CLINICAL TRIAL: NCT06852859
Title: Patient-reported Pain and Symptom Relief During Three Months After Surgery for Benign Prostatic Hyperplasia.
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Joakim Stromberg, Associate professor, Sahlgrenska University Hospital
Other Study IDs: 2024-06211-01 EPM
Record Dates: First submitted 2025-02-21; First posted 2025-02-28 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient treated by transurethral surgical procedure: Patients treated for BPH with surgery
  Interventions: Procedure: Transurethral resection of the prostate; Procedure: Transurethral vaporization of the prostate; Procedure: GreenLight laser enucleation of the prostate

INTERVENTIONS:
Procedure: Transurethral resection of the prostate — Thermocoagulation is used in contrast to the other methods
Procedure: Transurethral vaporization of the prostate — Heat is used to vaporize prostate
Procedure: GreenLight laser enucleation of the prostate — laser is used in contrast to the other methods

SUMMARY:
This is a prospective observational study in patients undergoing surgery for benign prostatic hyperplasia (BPH).

The purpose of the study is to investigate in great detail patients' recovery after surgery for BPH regarding pain, hematuria, urine leakage and use of pain-relieving medications for three months postoperatively. Patient-reported outcomes after three different surgical methods will be investigated: transurethral resection, transurethral vaporization and laser transurethral enucleation of the prostate (Green-LEP)

Research questions:

* How do patients rate their day-to-day pain during the first three months after surgery for BPH? How long does it take to be pain free?
* How does the patient estimate any day-to-day burning sensation during the first three months after surgery for BPH?
* How many painkilling tablets of a certain preparation and a certain strength take patients per day in the first three months after surgery for BPH?
* How long do patients have urinary leakage after surgery for BPH?
* Are the patients bothered by possible urine leakage and if so for how long after surgery for BPH?
* How long does one have macroscopic hematuria after surgery for BPH?
* How quickly are the patients' urinary tract problems affected according to the IPSS per month?
* Are the results on the above outcome measures different between the three TUR-P methods, TUV-P and Green LEP?

DETAILED DESCRIPTION:
Design and selection:

This is a prospective multicenter observational study in which patients undergoing TUR-P, TUV-P and GreenLEP for BPH are included. The subjects will be followed up with a self-assessment form that is completed daily for three months and then sent to the responsible researchers. After this, the research subjects will be followed up with sent out IPSS forms after six months, and then annually for up to five years. These are sent in stamped envelopes.

Participants:

The study will include 500 patients who undergo surgery for BPH at Alingsås hospital, Sjukhusen i Väster and Sahlgrenska University Hospital, as well as possibly an additional urology clinic in the future. The inclusion criteria include men over 50 years of age with diagnosed BPH and LUTS who have an indication for surgery with any of the three methods studied.

Outcome measures:

1. Pain and burning will be assessed using the NRS (numeric scale) between 0 and 10 where 0 is defined as "no pain/burning" and 10 is defined as "worst imaginable pain/burning". The researchers fill in this day-by-day for three months
2. Use of pain-relieving medications will be investigated with a table in which the research subjects enter drug names and sum up the number of tablets taken per day.
3. Urine leakage will be examined by the research subjects checking either "Yes" or "no" on the question of whether they have had urine leakage on a daily basis.
4. If this urine leakage has bothered the research subjects, it is investigated by ticking either "Yes" or "No" daily as a follow-up question to the previous one.
5. The duration of hematuria will be examined by the research subjects checking either "Yes" or "No" on the question of whether they have had blood in the urine daily
6. The change in LUTS measured by IPSS will be used to measure patient-perceived outcomes at baseline, after four, eight and twelve weeks, after six months and then annually for five years.

Data Analysis:

Descriptive statistics will be used to compile the PROMs data. Changes over time will be analyzed using repeated measures (ANOVA). Differences in outcome measures between the three different methods will be analyzed with the Mann-Whitney test for continuous, independent data pairs, and the Chi-Square test for categorical variables.

Ethical considerations:

The study will be conducted in accordance with the Declaration of Helsinki, and all participants will give their informed consent. Ethical approval will be sought from the Ethical Review Authority (EPM)

Significance and clinical relevance:

The results of this study will provide important insights into how patient-reported outcomes after benign prostate surgery can be used to improve surgical outcomes and patient counseling. The results will also be able to be used to compare outcome measures between the three different treatments used for BPH. By highlighting the patient's perspective, care can be developed to better meet the patients' needs and expectations, and by determining a "normal course" regarding these outcome measures, the results can also be used in the future to identify patients who deviate from the expected recovery course.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing transurethral surgery for benign prostatic hyperplasia
* Singed informed consent to participate

Exclusion Criteria:

* Non-swedish speaking patients

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery for benign prostatic hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative pain levels | Day-by-day for three months
  Day-by-day registration of pain by NRS (numeric response scale) for pain. Anchorpoints: 0 (no pain) to 10 (worst possible pain)

SECONDARY OUTCOMES:
Use of analgesics postoperatively | Day-by-day for three months
  Patients are to report all pain medication used day-by-day
Duration of postoperative hematuria | Day-by-day for three months
  The patients register the incidence of hematuria day-by-day by checking either "yes" or "no"
Duration of postoperative leakage of urine | Day-by-day for three months
  The patients record the incidence of leakage of urine day-by-day by checking either "yes" or "no" box
Concerns about urine leakage | Day-by-day for three months
  If the patients have checked the box "yes" for urine leakage, they are asked to record if they are bothered by this leakage or not by checking either "yes" or "no" box
Changes in Lower Urinary Tract Symptoms as measured by the IPSS questionnaire | Month-by-month for 3 months
  The patients are asked to complete the IPSS (International Prostatic Symptom Score) once a month. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Joakim BE Strömberg, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (3):
- Sweden (3):
  - Alingsås lasarett, department of general surgery, urology and orthopaedic surgery, Alingsås
  - Kungälvs sjukhus, department of urology, Kungälv
  - NU sjukvården, Uddevalla sjukhus, department of urology, Uddevalla

IPD SHARING:
Plan to Share IPD: Undecided